CLINICAL TRIAL: NCT06676943
Title: A Single Centre Pilot Study Investigating the Diagnostic Performance of High-resolution Specimen PET-CT in Determining Margin Status in Cancer Resection
Brief Title: Investigating the Diagnostic Performance of High-resolution Specimen PET-CT in Determining Margin Status in Cancer Resection
Acronym: eXcision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OA641624
Record Dates: First submitted 2024-10-31; First posted 2024-11-06 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer Surgery; Head and Neck Cancers
Keywords: specimen PET-CT; surgical margin status
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radical prostatectomy and Head and neck specimens (Experimental): Patients undergoing surgical resection for prostate cancer or head and neck cancer.
  Interventions: Procedure: XEOS AURA 10 specimen PET-CT scan of tumour specimens

INTERVENTIONS:
Procedure: XEOS AURA 10 specimen PET-CT scan of tumour specimens — Participants will be injected with a small amount of radioactive tracer at the beginning of their cancer operation. This tracer will attach itself to the cancer cells. Once the surgical specimen is removed it will be placed into the specimen PET-CT scanner so that the surgeon can see the cancer within the specimen and assess the margin.

SUMMARY:
Surgical removal is the treatment for many different cancers. Patient outcomes depend on complete cancer removal with no tumour present at the edge of the section removed (specimen). If cancer is left behind, then patients might need additional cancer treatment. Regardless of whether extra treatment is required, knowing that removal was incomplete causes anxiety. The need for a wide removal of the tumour must be balanced against the harm caused by more extensive surgery particularly when important organs and structures are close by. The fact that the cancer is not visible to the surgeon during the operation means that there is an element of guesswork when deciding how much tissue to remove. This study is examining a technique that the investigators hope will provide surgeons with more precise information about how much tissue to remove during cancer operations using a new type of Positron Emission Tomography-Computed Tomography (PET-CT) scanner. Patients with different types of cancer (e.g. prostate, head and neck cancer) will be injected with a small amount of radioactive tracer at the beginning of their cancer operation. This tracer will attach itself to the cancer cells. Once the surgical specimen is removed it will be placed into the specimen PET-CT scanner so that the surgeon can see the cancer within the specimen. The investigators will then compare the results of the scan of the specimen taken during the operation with the results when the whole specimen has been examined under the microscope. Examination under the microscope is considered to be the gold standard for deciding whether the cancer removal operation has been successful. This study aims to tell us how accurate the new specimen PET-CT scanner results are, and so whether or not surgeons can rely on the results to guide them during operations in the future.

ELIGIBILITY:
Inclusion Criteria:

For prostate cancer patients:

1. At least 18 years old at time of consent.
2. Listed for Robotic Radical Prostatectomy.

For head and neck cancer patients:

1. At least 18 years old at time of consent.
2. Listed for resection of oral squamous cell carcinoma head and neck cancer resection.
3. Specimen able to fit into Xeos Aura specimen container.

Exclusion Criteria:

For prostate cancer patients:

1. General or local contra-indications for resectional surgery.
2. Lacks capacity to provide informed consent.
3. Currently participating in another interventional research study that in the judgment of the investigator would negatively affect the participant and/or this study's data integrity.

For head and neck cancer patients:

1. General or local contra-indications for resectional surgery.
2. Lacks capacity to provide informed consent.
3. Pregnant or breast feeding patient.
4. Currently participating in another interventional research study that in the judgment of the investigator would negatively affect the participant and/or this study's data integrity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
To assess the accuracy of intra-operative high-resolution surgical specimen PET-CT (XEOS Aura 10) in determining margin status during prostate cancer resection, and head and neck cancer resection specimens compared to the reference gold standard. | Up to 8 weeks after the day of surgery when the histopathological margin status result is recorded.
  The true gold standard is whether the cancer is on the margin (positive) or not (negative) as per specimen PET-CT compared to the gold standard radical prostatectomy histopathological margin status, and head and neck cancer resection specimen.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Coventry and Warwickshire NHS Trust, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided